CLINICAL TRIAL: NCT06315946
Title: Prospective, Single-blinded, Randomized Trial to Evaluate the Efficacy of a Cryogenic Medical Device on Skin Tags Versus a Comparator Product.
Brief Title: Efficacy of a Cryogenic Medical Device on Skin Tags Versus a Comparator Product.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17E3241
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Skin Tags

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pixie® skin tag (Experimental): A skin tag is selected and treated with the test device Pixie® skin tag according to the instructions for use.
  Interventions: Device: Pixie® skin tag
- Wortie® skin tag remover (Active Comparator): A skin tag is selected and treated with the comparator Wortie® skin tag remover.
  Interventions: Device: Wortie® Skin Tag Remover

INTERVENTIONS:
Device: Pixie® skin tag — The skin tag is treated by treatment with the cryogenic device. To protect the surrounding skin, a protective foam plaster is applied before the device is used on the skin tag. The skin tag is treated for 20 seconds after loading the device for 2 seconds.
  Arms: Pixie® skin tag
Device: Wortie® Skin Tag Remover — The skin tag is treated by treatment with the cryogenic device. The frozen metal nib is applied on the skin tag for 40 seconds.
  Arms: Wortie® skin tag remover

SUMMARY:
Evaluate the efficacy of the test medical device (Pixie® skin tag) in the treatment of skin tags versus a comparator product (Wortie® skin tag remover).

DETAILED DESCRIPTION:
The main objective of the study was to evaluate the efficacy of the test medical device Pixie® skin tag) in the treatment of skin tags versus a comparator product (Wortie® skin tag remover). Non-inferiority of the test product versus competitor on skin tag evaluated by clinical evaluation.

The secondary objectives of the study were to evaluate:

* the number of treatments needed for the complete disappearance of skin tag;
* the efficacy of devices by subjects' self-assessment;
* the cutaneous tolerability (safety).

The last objective of the study was to illustrate the expected visual effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject
* Sex: male or female
* Age: between 18 and 65 years old
* Type: Caucasion
* Phototype: I to III according to Fitzpatrick
* Subject presenting at least one skin tag that could be treated by the tested devices on the neck, the breast, or under armpits of 2 to 5 mm diameter.
* Subject having given freely and expressly his/her informed consent.
* Subject who is able to comply with the study requirements, as defined in the present CIP, at the investigator's appreciation.
* Subject being affiliated to a health social security system.
* Female subjects of childbearing potential should use a medically accepted contraceptive regimen since at least 4 weeks before the beginning of the study and during all the study.

Exclusion Criteria:

* Pregnant, parturient, nursing woman or woman planning a pregnancy during the study.
* Subject who had been deprived of their freedom by administrative or legal decision.
* Subject who is under guardianship.
* Subject having received 4500 euros indemnities for participation in clinical trials in the 12 previous months, including participation in the present study.
* Subject currently participating in another research or being in an exclusion period for a previous study.
* Subject suffering from an acute disease or any other pathology that may interfere with the evaluation of the study results at the investigator's opinion.
* Subject with a cutaneous disease that may interfere with the evaluation of the study results or might put the subject at undue risk at the investigator's opinion.
* Subject with a history of skin cancer.
* Subject with a history of pre-cancerous skin lesions.
* Subject with a known allergy to one of the component of the products, to the comparator, to nickel, to Biseptine® or any other Chlorhexidine based antiseptic or to the adhesive.
* Subject suffering from asthma.
* Subject who has diabetes.
* Subject with previous event of healing disorders as hypertrophic or keloid scar, residual pigmentation etc.
* Subject with blood circulation or blood clotting problems including Raynaud's disease; blood dyscrasias of unknown origin; haemophilia subjects.
* Subject with immune deficiency or autoimmune disease.
* Subject presenting birthmarks, moles, warts, or any other spots on the studied zone.
* Subject having an inflamed, infected, irritated, red, damaged, cut, grazed, diseased or itchy skin on the treated zone.
* Subject who already had an abnormal reaction to cold.
* Subject whose selected skin tag is bleeding or scratched.
* Subject undergoing a topical treatment on the test area or a systemic treatment:
* anti-inflammatory medication during the previous 5 days and during the study,
* immunosuppressors and/or corticoids during the 10 previous days and during the study,
* retinoids during the 6 previous months and during the study,
* treatment with an action on coagulation during the previous week and during the study,
* any long-term medication stabilized for less than one month.
* Subject who received a treatment of any type on the selected skin tag during the previous 6 months.
* Intensive exposure to sunlight or UV-rays within the previous month and/or foreseen exposure of the treated zone during the study.
* Subject planning to change her/his life habits during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with successful treatment | day 45 +-2 days
  Comparison of the percentage of subjects having a successful treatment of their skin tag in the test group versus the comparator; clinical evaluation by a blinded evaluator.

SECONDARY OUTCOMES:
Number of treatments | day 45 +-2 days
  Comparison of the number of treatments needed for clinical remission of the skin tag with both products, as assessed by the blinded evaluator.
Visual aspect | Every day (for a period of 45 days +- 2 days)
  Evaluation of devices efficacy by subjects' self-assessment, using a subjective evaluation questionnaire completed at the study end.
Macrophotographs on skin tag remission | Day 0 (before treatment); day 15 (before treatment); day 30 (before treatment) and day 45 if applicable.
  Illustration of the visual aspects of the process of skin tag remission by realisation of macrophotographs.
Evaluation of the skin condition | Day 0, Day 3 (+-1day), Day 15 (+-2days), Day 30 (+-2days) and Day 45(+-2days)
  Evaluation of the skin conditions to assess products tolerability at each timepoint, assessed by the investigator by clinical evaluation.
Degree of pain | During treatement on day 0, and if applicable on follow-up treatments on day 15 and day 30.
  Evaluation of the degree of pain felt by subjects during the treatment.
Recording of adverse events | Day 0, Day 3 (+-1day), Day 15 (+-2days), Day 30 (+-2days) and Day 45(+-2days)
  Recording of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Bathelier, PhD, Principal Investigator — Dermscan/Pharmascan
Locations (1):
- DERMSCAN - PharmScan, Villeurbanne, France